CLINICAL TRIAL: NCT03801057
Title: The Effect of a Marine Protein Hydrolysate Supplement on Inflammatory Markers, Microbiota Composition and Symptoms in Patients With Irritable Bowel Syndrome
Brief Title: Marine Protein Hydrolysate as Dietary Supplement in Irritable Bowel Syndrome
Acronym: MPH_IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Haukeland University Hospital (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/1825
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Dietary Supplements; Fish Proteins; Protein Hydrolysates
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: A parallel group randomized, controlled clinical trial for six weeks
Who Masked: Participant, Care Provider, Investigator
Masking Description: The provider of the dietary supplement deliver the supplement prepared and packed in equal bags (active/placebo) that we hand out to the participants in an randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPH_active (Active Comparator): Daily intake at breakfast of supplementary marine protein hydrolysate (MPH). Random sequence of arms.
  Interventions: Dietary Supplement: MPH_active
- MPH_placebo (Placebo Comparator): Daily intake at breakfast of supplementary placebo. Random sequence of arms.
  Interventions: Dietary Supplement: MPH_placebo

INTERVENTIONS:
Dietary Supplement: MPH_active — One daily intake at breakfast of supplementary marine protein hydrolysate (MPH), a dosage of 2400 mg, duration 6 weeks. The form is powder, flavored with lemon, and to be mixed with 100 ml water. Random sequence of arms.
  Arms: MPH_active
Dietary Supplement: MPH_placebo — One daily intake at breakfast of supplementary placebo, a dosage of 2400 mg, duration 6 weeks. The form is powder, flavored with lemon, and to be mixed with 100 ml water.
  Arms: MPH_placebo

SUMMARY:
The use of natural bioactive products for prevention and treatment of a wide spectrum of conditions, including gastrointestinal disorders and conditions is well known. Based on current evidences, the scientific validity of such products is limited. However, there is sufficient preliminary data to indicate that bioactive compounds may be novel for potentially clinical use, thus further clinical trials investigating effect are needed. This trial is meant to evaluate the effect of an marine protein hydrolysate (MPH) supplement on composition of microbiota, inflammatory markers and symptom severity in people diagnosed with irritable bowel syndrome.

DETAILED DESCRIPTION:
Previous studies performed in rodents have found that hydrolyzed proteins from fish alters the lipid and cholesterol metabolism, reduce plasma cholesterol and triglyceride levels and alters the fatty acid composition in liver and adipose tissue. Previous studies in humans have found marine peptides to have both antihypertensive and antioxidant effects. It is also suggested that fish protein hydrolysates may have an immunomodulating effect with beneficial properties in the intestine, and may prevent NSAID-induced injuries, change permeability in the gut and possibly prevent injurious conditions in the gut.

The evidence and knowledge are limited on the interaction between diet, gut microbiota and the influence of specific nutrients, as well as the impact of different sources of proteins on inflammation markers, gut microbiota and symptom severity in patients with irritable bowel syndrome (IBS). Different dietary sources of protein affect the diversity and composition of the human gut microbiota in different degree, demonstrated by a distinct gut bacteria profile observed between omnivores and vegetarians.The specific effect of marine peptides on human gut microbiota composition is as far as the investigators know, previously not investigated. Interestingly, novel results indicate that the presence of fish proteins in the diet have impact on both composition and activity of the gut microbiome, influencing the human microbiota composition.

The many benefits of expanding the utilization of marine products, the previous assumed beneficial intestinal effect and the increased interest in gut health and microbiota, as well as a great need for novel dietary treatment strategies for patients with irritable bowel syndrome (IBS) make this study warrant.

Aim with this trial is to evaluate the effect of an marine protein hydrolysate (MPH) supplement on composition of microbiota, inflammatory markers and symptom severity in human subjects diagnosed with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) 18-30 kg/m2
* Irritable Bowel Syndrome (IBS) diagnosis according to Rome IV criteria

Exclusion Criteria:

* Suspected allergies against fish or shellfish
* Low or unstable blood pressure
* Diabetes mellitus pharmacologically treated
* Chronic diseases or therapies that are likely to interfere with the evaluation of study results such as known inflammation
* Acute infections (may be reconsidered for inclusion at a later time)
* Substance misuse
* Inability or unwillingness to comply with the requirements of study procedures
* Individuals in the middle of testing different dietary strategies for the treatment of IBS (such as the low-FODMAP diet) and/or not willing to/able to maintain a stable diet throughout the study period
* Use of pro- or prebiotic supplements
* Use of antibiotic treatment for the last 4 weeks
* Immunocompromised patient defined as taking immuno-suppressive medications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
IBS-SSS | Before (baseline) and after intervention (6 weeks later).
  A decrease of 50 points or more in IBS-SSS, which is a clinically meaningful improvement.The IBS-SSS is a 5-question survey that asks the severity of abdominal pain, frequency of abdominal pain, severity of abdominal distention, dissatisfaction with bowel habits, and interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Scores on the IBS-SSS can range from 0 to 500 with higher scores indicating more severe symptoms. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS.

SECONDARY OUTCOMES:
SF-NDI_HRQOL | Before (baseline) and after intervention (6 weeks later).
  The Short Form (SF) Nepean Dyspepsia Index is a 10-item questionnaire with 5 sub-scales each examining the influence of dyspepsia on domains of health in patients, namely tension/anxiety, interference with daily activities, disruption to regular eating/drinking, knowledge towards/control over disease symptoms and interference with work/study, with each sub-scale containing two items . Each item is measured by a 5-point Likert scale ranging from 0 (not at all or not applicable), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely). Individual items in each sub-scale are aggregated to obtain a score range from 0 (lowest HRQoL score) to 100 (highest HRQoL score) as per the developers' original calculation formula. A total, overall SF-NDI total score is obtained using the mean of 5 subscale scores.
Fecal Calprotectin | Before (baseline) and after intervention (6 weeks later).
  Calprotectin is a protein found in several human fluids. When detected in the stool, calprotectin has a direct relationship (consequence of neutrophil degranulation) to inflammation in the bowel.

OTHER OUTCOMES:
Inflammatory markers in blood | Before (baseline) and after intervention (6 weeks later).
  Zonulin, iFABP (intestinal fatty acid binding protein), LBP (lipopolysaccharide binding protein), IL-4, 6, 8, 10, TNF-α and INF-γ are markers of bowel mucosal damage.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne Lihaug Hoff, MD, PhD, Study Director — Helse Møre og Romsdal Hospital Trust
Locations (2):
- Norway (2):
  - Ålesund Hospital, Helse Møre og Romsdal HF, Ålesund
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dale HF, Jensen C, Hausken T, Valeur J, Hoff DAL, Lied GA. Effects of a Cod Protein Hydrolysate Supplement on Symptoms, Gut Integrity Markers and Fecal Fermentation in Patients with Irritable Bowel Syndrome. Nutrients. 2019 Jul 17;11(7):1635. doi: 10.3390/nu11071635. PMID 31319590